CLINICAL TRIAL: NCT02326025
Title: An Open-Label Study to Evaluate the Pharmacokinetics of Doxorubicin Following the Concomitant Intravenous Administration of Olaratumab (IMC-3G3) to Patients With Advanced Soft Tissue Sarcoma
Brief Title: A Study of Olaratumab and Doxorubicin in Participants With Advanced Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 15676; I5B-EW-JGDI (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-12-22; First posted 2014-12-25 (Estimated); Results first posted 2019-11-21 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-04

CONDITIONS: Sarcoma, Soft Tissue
MeSH Terms: conditions — Sarcoma | interventions — olaratumab; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part A (Experimental): Doxorubicin Alone: On Cycle 1, Day 1, participants received 75 milligram/square meter (mg/m2) of doxorubicin intravenously (IV).
  Olaratumab Alone: On Cycle 1, Day 10, participants received 15 milligram/kilogram (mg/kg) of olaratumab IV.
  Olaratumab + Doxorubicin: For Cycles 2 to 8, participants received 15 mg/kg of olaratumab on Days 1 and 8 of each 21-day cycle, IV and 75 mg/m2 of doxorubicin IV immediately following the completion of the olaratumab infusion.
  Participants continued to receive olaratumab monotherapy (on days 1 and 8 of each cycle) for Cycle 9 onward, until discontinuation criteria are met.
  Interventions: Drug: Olaratumab; Drug: Doxorubicin
- Part B (Experimental): Doxorubicin Alone: On Cycle 1, Day 1, participants received doxorubicin 75 mg/m2 IV
  Olaratumab Alone: On Cycle 1, Day 10, participants received 20 mg/kg of olaratumab IV.
  Olaratumab + Doxorubicin:
  For Cycle 2, participants received 20 mg of olaratumab on Days 1 and 8 of each 21-day cycle, IV. On Day 1 of Cycle 2, doxorubicin 75 mg/m2 was administered IV immediately following the completion of the olaratumab infusion.
  For Cycles 3 - 8, Day 1 and 8, olaratumab 15 mg/kg was administered and on Day 1 doxorubicin 75 mg/m2 was administered IV immediately following the completion of the olaratumab infusion.
  Participants continued to receive olaratumab monotherapy (on days 1 and 8 of each cycle) for Cycle 9 onwards, until discontinuation criteria are met.
  Interventions: Drug: Olaratumab; Drug: Doxorubicin

INTERVENTIONS:
Drug: Olaratumab — Administered IV
  Other Names: LY3012207; IMC-3G3
Drug: Doxorubicin — Administered IV

SUMMARY:
The purpose of this study is to assess how the body handles olaratumab when it is given with another drug called doxorubicin.

The safety and tolerability of these drugs will be studied. Each participant will complete two 21-day cycles in a fixed order. Participants who complete Cycle 2 may continue to receive olaratumab + doxorubicin for an additional six 21-day cycles and then may receive olaratumab alone until discontinuation criteria are met.

Screening is required within 21 days prior to first dose.

Part B was added in October, 2015 to assess how the body handles a higher dose of olaratumab when given with doxorubicin.

Participants may only enroll in one part.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of soft tissue sarcoma (STS) that is advanced and/or metastatic
* Have the presence of measurable and/or nonmeasurable disease
* Have given written informed consent prior to any study-specific procedures
* Have a performance status of less than or equal to 2 on the Eastern Cooperative Oncology Group (ECOG) scale
* Have discontinued previous treatments for cancer and recovered from the acute effects of therapy
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures

Exclusion Criteria:

* Have received treatment within 28 days of the initial dose of study drug with an investigational product or non-approved use of a drug or device for noncancer indications
* Have received prior treatment with doxorubicin, daunorubicin, idarubicin, and/or other anthracyclines and anthracenediones
* Have active central nervous system (CNS) metastasis. Participants with treated CNS metastases are eligible for this study if they are not currently receiving corticosteroids
* Have unstable hepatic disease with a grade equal to or greater than Child-Pugh B
* Have an active fungal, bacterial, and/or known viral infection including human immunodeficiency virus (HIV) or viral (A, B, or C) hepatitis
* Have a history of another primary cancer, with the exception of a) curatively resected nonmelanoma skin cancer; b) curatively treated cervical carcinoma in situ; or c) other primary solid tumor treated with curative intent, no known active disease present, and no treatment administered during the last 3 years prior to study entry
* Have a history of chronic heart failure or left ventricular dysfunction
* Have a resting heart rate of less than (<)50 beats per minute (bpm) or greater than (>)100 bpm
* Have a history of radiation therapy involving the mediastinal/pericardial area. Previous radiation therapy is allowed but must not have included whole pelvis radiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2015-05-20 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (6):
- United States (6):
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - IU Simon Cancer Center, Indianapolis, Indiana
  - Washington University Medical Center, St Louis, Missouri
  - Seattle Cancer Care Alliance, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Completers include participants who died or discontinued study treatment due to progressive disease.
Groups:
- Part A: Doxorubicin (Dox) Alone: On Cycle 1, Day 1, participants received 75 milligram/square meter (mg/m2) of doxorubicin intravenously (IV).
  Olaratumab Alone: On Cycle 1, Day 10, participants received 15 milligram/kilogram (mg/kg) of olaratumab IV.
  Olaratumab + Doxorubicin: For Cycles 2 to 8, participants received 15 mg/kg of olaratumab on Days 1 and 8 of each 21-day cycle, IV and 75 mg/m2 of doxorubicin IV immediately following the completion of the olaratumab infusion.
  Participants continued to receive olaratumab monotherapy (on days 1 and 8 of each cycle) for Cycle 9 onward, until discontinuation criteria are met.
Period: Overall Study
Arm/Group | Part A | Part B
Started | 25 | 24
Received at Least 1 Dose of Study Drug | 25 | 24
Completed | 20 | 19
Not Completed | 5 | 5
Not completed — Adverse Event | 3 | 0
Not completed — Physician Decision | 1 | 2
Not completed — Physician and Participant Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A | Part B | Total
Number analyzed (Participants) | 25 | 24 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (12.6) | 56.1 (11.2) | 56.4 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 14 | 29
  Male | 10 | 10 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 24 | 22 | 46
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 1 | 4
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 24 | 49

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Area Under The Concentration Curve Zero to Infinity (AUC[0-∞]) Doxorubicin
Time Frame: Cycle(C)1 and (C)2, Day(D)1: Predose, 0.5, 1, 2, 4, 8, 24, 48, 72, 96 Hours (Hrs) Post dose
Population: All participants who received at least one dose of study drugs and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour/milliliter (ng*h/mL)
Groups:
- Part A Doxorubicin Alone; Part B Doxorubicin Alone: On Cycle 1, Day 1, participants received 75 milligram/square meter (mg/m2) of doxorubicin IV.
- Part A Doxorubicin + 15 mg/kg Olaratumab: On Cycle 1, Day 1, participants received 75 mg/m2 of doxorubicin IV and then on Cycle 1, Day 1, participants received 15 milligram/kilogram (mg/kg) of olaratumab IV.
- Part B Doxorubicin + 20 mg/kg Olaratumab: On Cycle 2, Day 1, participants received 75 mg/m2 of doxorubicin IV immediately following the completion of the 20 mg/kg of olaratumab infusion.
Arm/Group | Part A Doxorubicin Alone | Part A Doxorubicin + 15 mg/kg Olaratumab | Part B Doxorubicin Alone | Part B Doxorubicin + 20 mg/kg Olaratumab
Number analyzed (Participants) | 23 | 22 | 24 | 21
nanogram*hour/milliliter (ng*h/mL) | 2580 (24) | 2570 (28) | 2400 (21) | 2470 (20)
Statistical Analysis 1: Comparison: Part A Doxorubicin Alone vs Part A Doxorubicin + 15 mg/kg Olaratumab; Test type: Superiority; Ratio of Geometric LS Means = 1.04, 90% CI 2-sided [0.964 to 1.13] — Log(PK) is participant and treatment and random error, where participant is fitted as a random effect
Statistical Analysis 2: Comparison: Part B Doxorubicin Alone vs Part B Doxorubicin + 20 mg/kg Olaratumab; Test type: Superiority; Ratio of LS Means = 1.03, 90% CI 2-sided [0.957 to 1.11]

2. Primary Outcome: PK: Maximum Concentration (Cmax) Doxorubicin
Time Frame: C1 and C2, D1: Predose, 0.5, 1, 2, 4, 8, 24, 48, 72, 96 Hrs Post dose
Population: All participants who received at least one dose of study drugs and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/ml)
Groups:
- Part A Doxorubicin Alone: On Cycle 1, Day 1, participants received 75 mg/m2 of doxorubicin, IV.
Arm/Group | Part A Doxorubicin Alone | Part A Doxorubicin + 15 mg/kg Olaratumab | Part B Doxorubicin Alone | Part B Doxorubicin + 20 mg/kg Olaratumab
Number analyzed (Participants) | 23 | 22 | 24 | 21
nanogram/milliliter (ng/ml) | 2570 (47) | 2330 (68) | 2060 (53) | 2070 (60)
Statistical Analysis 1: Comparison: Part A Doxorubicin Alone vs Part A Doxorubicin + 15 mg/kg Olaratumab; Test type: Superiority; Ratio of LS Means = 0.944, 90% CI 2-sided [0.770 to 1.16]
Statistical Analysis 2: Comparison: Part B Doxorubicin Alone vs Part B Doxorubicin + 20 mg/kg Olaratumab; Test type: Superiority; Ratio of LS Means = 1.03, 90% CI 2-sided [0.801 to 1.33]

3. Secondary Outcome: PK:Time of Maximum Observed Concentration (Tmax) Doxorubicin
Time Frame: C1 and C2, D1: Predose, 0.5, 1, 2, 4, 8, 24, 48, 72, 96 Hrs Post dose
Population: All participants who received at least one dose of study drugs and had evaluable PK data.
Measure: Median (Full Range); unit: hour (h)
Arm/Group | Part A Doxorubicin Alone | Part A Doxorubicin + 15 mg/kg Olaratumab | Part B Doxorubicin Alone | Part B Doxorubicin + 20 mg/kg Olaratumab
Number analyzed (Participants) | 23 | 22 | 24 | 21
hour (h) | 0.30 [0.25 to 0.58] | 0.31 [0.25 to 0.58] | 0.33 [0.25 to 0.67] | 0.33 [0.25 to 0.55]

4. Secondary Outcome: PK: AUC Zero to Time t, Where t is the Last Time Point (0-tLast) Olaratumab
Description: PK: AUC (0-tLast) with a measurable concentration. PK data includes Part A Olaratumab alone and Part B Olaratumab + Doxorubicin.
Time Frame: C1 D10: Predose, 0, 1, 4, 24, 48, 72, 96 Hrs Post dose; C2 D1: Predose, 0, 1, 4, 24, 48, 72, 96 Hrs Post dose
Population: All participants who received at least one dose of study drugs and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng∙h/mL
Groups:
- Olaratumab Alone Part A: On Cycle 1, Day 1, participants received 75 milligram/square meter (mg/m2) of doxorubicin IV.
- Part A 15 mg/kg Olaratumab + Doxorubicin: On Cycle 1, Day 1, participants received 75 mg/m2 of doxorubicin IV and then on Cycle 1, Day 10, participants received 15 milligram/kilogram (mg/kg) of olaratumab IV.
- Part B Olaratumab Alone: On Cycle 1, Day 10, participants received 20 mg/kg of olaratumab, IV
- Part B 20 mg/kg Olaratumab + Doxorubicin: On Cycle 2, Day 1, participants received 75 mg/m2 of doxorubicin IV immediately following the completion of the 20 mg/kg of olaratumab infusion.
Arm/Group | Olaratumab Alone Part A | Part A 15 mg/kg Olaratumab + Doxorubicin | Part B Olaratumab Alone | Part B 20 mg/kg Olaratumab + Doxorubicin
Number analyzed (Participants) | 23 | 24 | 23 | 23
ng∙h/mL | 32800 (21) | 32000 (21) | 53800 (24) | 54100 (20)

5. Secondary Outcome: PK: Cmax Olaratumab
Description: PK data includes Part A Olaratumab alone and Part B Olaratumab + Doxorubicin.
Time Frame: C1 D10:Predose, 0, 1, 4, 24, 48, 72, 96 Hrs Post dose; C2 D1: Predose, 0, 1, 4, 24, 48, 72, 96 Hrs Post dose
Population: All participants who received at least one dose of study drugs and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Part A Olaratumab Alone: On Cycle 1, Day 10, participants received 15 mg/kg of olaratumab, IV.
Arm/Group | Part A Olaratumab Alone | Part A 15 mg/kg Olaratumab + Doxorubicin | Part B Olaratumab Alone | Part B 20 mg/kg Olaratumab + Doxorubicin
Number analyzed (Participants) | 23 | 24 | 23 | 23
ng/mL | 292 (19) | 386 (16) | 512 (21) | 634 (26)

6. Secondary Outcome: PK: Tmax Olaratumab
Description: Tmax times are relative to the start of the approximately 60-minute IV infusion of olaratumab. PK data includes Part A Olaratumab alone and Part B Olaratumab + Doxorubicin.
Time Frame: C1 D10: Predose, 0, 1, 4, 24, 48, 72, 96 Hrs Post dose; C2 D1: Predose, 0, 1, 4, 24, 48, 72, 96 Hrs Post dose
Population: All participants who received at least one dose of study drugs and had evaluable PK data.
Measure: Median (Full Range); unit: h
Arm/Group | Part A Olaratumab Alone | Part A 15 mg/kg Olaratumab + Doxorubicin | Part B Olaratumab Alone | Part B 20 mg/kg Olaratumab + Doxorubicin
Number analyzed (Participants) | 23 | 24 | 23 | 23
h | 2.00 [1.00 to 23.17] | 2.79 [1.80 to 6.43] | 1.67 [0.05 to 24.10] | 3.50 [1.00 to 6.97]

7. Secondary Outcome: Percentage of Participants With Olaratumab Antibodies
Description: The formation of anti-drug antibodies (ADA) was assessed using validated ELISAs, following a 4-tier approach. Both the ADA screening assay and the neutralizing antibody assay were validated in accordance with the US Food and Drug Administration (FDA) Guidance for Industry. Participants who had positive samples for treatment emergence due to being <4-fold difference from baseline or occurred prior to drug exposure are reported.
Time Frame: Preinfusion on Day 1 of Cycles 1 through 3 and Preinfusion on Day 1 of Every Second Cycle Thereafter, Up to 30-Day Follow Up
Population: All participants who received at least one dose of study drug and had evaluable baseline and post-baseline anti-olaratumab antibodies.
Measure: Number; unit: percentage of participants
Groups:
- Part A 15 mg/kg Olaratumab: Olaratumab Alone: On Cycle 1, Day 10, participants received 15 milligram/kilogram (mg/kg) of olaratumab IV.
  Participants continued to receive olaratumab monotherapy (on days 1 and 8 of each cycle) for Cycle 9 onward, until discontinuation criteria are met.
- Part B 20 mg/kg Olaratumab: Olaratumab Alone: On Cycle 1, Day 10, participants received 20 mg/kg of olaratumab IV.
  Participants continued to receive olaratumab monotherapy (on days 1 and 8 of each cycle) for Cycle 9 onwards, until discontinuation criteria are met.
Arm/Group | Part A 15 mg/kg Olaratumab | Part B 20 mg/kg Olaratumab
Number analyzed (Participants) | 25 | 24
percentage of participants | 0 | 0

8. Secondary Outcome: Percentage of Participants With a Best Overall Response of Complete Response (CR) or Partial Response (PR) [Objective Response Rate (ORR)]
Description: The percentage of participants with a best overall response achieving CR or PR (ORR) was defined using Response Evaluation Criteria In Solid Tumors (RECIST, version 1.1) criteria. Complete Response (CR) was defined as the disappearance of all target and non-target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeter (mm) and normalization of tumor marker level of non-target lesions; Partial Response (PR) was defined as having at least a 30% decrease in sum of longest diameter of target lesions. The methodology for the confidence interval calculation is the "exact F" method.
Time Frame: Baseline to Measured Progressive Disease, Study Discontinuation or Death (Up to 24 Months)
Population: All participants who received at least one dose of study drug and had a post-baseline lesion response.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part A Dox Alone, Then Olaratumab Alone, Then Dox + Olaratumab: Doxorubicin Alone: On Cycle 1, Day 1, participants received 75 milligram/square meter (mg/m2) of doxorubicin intravenously (IV).
  Olaratumab Alone: On Cycle 1, Day 10, participants received 15 milligram/kilogram (mg/kg) of olaratumab IV.
  Olaratumab + Doxorubicin: For Cycles 2 to 8, participants received 15 mg/kg of olaratumab on Days 1 and 8 of each 21-day cycle, IV and 75 mg/m2 of doxorubicin IV immediately following the completion of the olaratumab infusion.
  Participants continued to receive olaratumab monotherapy (on days 1 and 8 of each cycle) for Cycle 9 onward, until discontinuation criteria are met.
- Part B Dox Alone, Then Olaratumab Alone, Then Dox + Olaratumab: Doxorubicin Alone: On Cycle 1, Day 1, participants received doxorubicin 75 mg/m2 IV
  Olaratumab Alone: On Cycle 1, Day 10, participants received 20 mg/kg of olaratumab IV.
  Olaratumab + Doxorubicin:
  For Cycle 2, participants received 20 mg of olaratumab on Days 1 and 8 of each 21-day cycle, IV. On Day 1 of Cycle 2, doxorubicin 75 mg/m2 was administered IV immediately following the completion of the olaratumab infusion.
  For Cycles 3 - 8, Day 1 and 8, olaratumab 15 mg/kg was administered and on Day 1 doxorubicin 75 mg/m2 was administered IV immediately following the completion of the olaratumab infusion.
  Participants continued to receive olaratumab monotherapy (on days 1 and 8 of each cycle) for Cycle 9 onwards, until discontinuation criteria are met.
Arm/Group | Part A Dox Alone, Then Olaratumab Alone, Then Dox + Olaratumab | Part B Dox Alone, Then Olaratumab Alone, Then Dox + Olaratumab
Number analyzed (Participants) | 25 | 24
percentage of participants | 12.0 [2.5 to 31.2] | 25.0 [9.8 to 46.7]

ADVERSE EVENTS:
Time Frame: From Baseline, to Study Completion (Up to 47 Months)
Description: All participants in the safety population received at least 1 dose of study drug and at least 1 post dose safety assessment.
Arm/Group | Part A | Part B
Serious Adverse Events (participants affected / at risk) | 9/25 | 9/24
Other Adverse Events (participants affected / at risk) | 24/25 | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=25) | Part B (N=24)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis salmonella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1)
Embolism venous (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A (N=25) | Part B (N=24)
Anaemia (Blood and lymphatic system disorders) | 10 (11) | 8 (10)
Neutropenia (Blood and lymphatic system disorders) | 9 (12) | 7 (10)
Thrombocytopenia (Blood and lymphatic system disorders) | 7 (11) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Dry eye (Eye disorders) | 2 (4) | 1 (1)
Eye pain (Eye disorders) | 2 (2) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 6 (7)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 9 (9) | 12 (20)
Diarrhoea (Gastrointestinal disorders) | 6 (7) | 12 (22)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 7 (7)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 (7) | 3 (6)
Nausea (Gastrointestinal disorders) | 13 (14) | 19 (31)
Stomatitis (Gastrointestinal disorders) | 5 (6) | 4 (4)
Vomiting (Gastrointestinal disorders) | 5 (6) | 8 (14)
Asthenia (General disorders) | 2 (2) | 1 (1)
Chills (General disorders) | 3 (3) | 1 (1)
Fatigue (General disorders) | 14 (19) | 18 (24)
Mucosal inflammation (General disorders) | 3 (4) | 8 (10)
Non-cardiac chest pain (General disorders) | 1 (1) | 3 (3)
Oedema (General disorders) | 2 (2) | 1 (1)
Oedema peripheral (General disorders) | 2 (2) | 5 (5)
Pyrexia (General disorders) | 2 (2) | 4 (6)
Temperature intolerance (General disorders) | 0 (0) | 2 (2)
Candida infection (Infections and infestations) | 0 (0) | 2 (2)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Oral candidiasis (Infections and infestations) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 5 (8)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (3)
Activated partial thromboplastin time prolonged (Investigations) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 0 (0) | 3 (4)
Ejection fraction decreased (Investigations) | 2 (2) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 3 (3)
International normalised ratio increased (Investigations) | 1 (1) | 2 (2)
Lymphocyte count decreased (Investigations) | 4 (4) | 1 (3)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (7)
Platelet count decreased (Investigations) | 3 (4) | 2 (10)
Weight decreased (Investigations) | 2 (2) | 2 (2)
White blood cell count decreased (Investigations) | 6 (8) | 4 (9)
Decreased appetite (Metabolism and nutrition disorders) | 7 (7) | 8 (9)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (9)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (3)
Dizziness (Nervous system disorders) | 4 (5) | 7 (10)
Dysgeusia (Nervous system disorders) | 4 (6) | 8 (9)
Headache (Nervous system disorders) | 6 (6) | 4 (4)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (2) | 3 (4)
Depression (Psychiatric disorders) | 2 (2) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 3 (3)
Dysuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 2 (2)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (8)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (4)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (7)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 7 (7) | 10 (10)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Nail discolouration (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3)
Embolism (Vascular disorders) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 3 (3)
Hypotension (Vascular disorders) | 0 (0) | 2 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days